CLINICAL TRIAL: NCT01873196
Title: Food Aid Quality Review: Feasibility and Acceptability Study of Corn Soy Blend and Fortified Vegetable Oil in Malawi
Acronym: FAQR-Malawi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: AID-016-Malawi; AFP-C-00-09-00016-00 (Other Grant/Funding Number: USAID)
Record Dates: First submitted 2013-04-22; First posted 2013-06-10 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Child Malnutrition
MeSH Terms: conditions — Child Nutrition Disorders

ARMS (4):
- Receive extra oil (Experimental): This arm will receive enough oil to prepare the CSB they receive in the newly recommended proportion of 100g CSB: 30g oil. They will receive education and instructions on the new method of preparation.
  Interventions: Behavioral: Receive extra oil
- Control-No extra oil received (No Intervention): This group will continue to receive only 1L of oil with their CSB has they already have been. They also will not receive any new education.
- Receives behavior changed messages on CSB package (Experimental): Group receiving CSB repackaged into 2kg packages with messages on package on how to prepare. Only in Phase II.
  Interventions: Behavioral: Receives behavior changed messages on CSB package
- Control-No repackaged CSB (No Intervention)

INTERVENTIONS:
Behavioral: Receive extra oil
  Arms: Receive extra oil
Behavioral: Receives behavior changed messages on CSB package
  Arms: Receives behavior changed messages on CSB package

SUMMARY:
This research will test alternative methods of ensuring compliance with recommended preparation and targeting of supplementary foods for malnourished children under five years of age.

The hypotheses that the proposed study intends to test are as follows:

1. With appropriate behavior change communication (BCC) and social support, and with provision of CSB and FVO in the correct proportions, it is possible to get women to prepare CSB with oil in the recommended ratio of 100:30, and in quantities just sufficient for the target child.
2. Providing CSB to Beneficiary Mothers/Caretakers pre-packaged bags of 2 kg with appropriate messaging and with instructions to direct the food to children and to prepare the CSB with oil in the recommended ratio and feed as instructed will result in better compliance.

DETAILED DESCRIPTION:
The first stage of the study involves working with the procurement and program staff to ensure that oil and CSB will be available at the same time in sufficient quantities and can be distributed together. We will work with program staff and outside consultants (if needed) to develop locally acceptable recipes for CSB plus oil. A sample of communities with MCHN programs will be chosen, and the intervention (consistent provision of CSB with oil, teaching of recipes using CSB with oil, appropriate behavioral support) implemented. Tufts and locally contracted researchers will interview program staff involved in procurement and supply chain management as well as program staff, and beneficiaries, to assess the feasibility and acceptability of the provision of CSB with oil, and identify barriers and problems. This stage is expected to take six months.

In the second stage of the study, the CSB will be distributed in new, smaller packages in half the sample communities, with the other half continuing with their normal distribution. In preparation for this stage, during the first stage, Tufts researchers will arrange for the production/packaging of a sufficient supply of CSB in the new packages, and will contract with local communications specialists to develop appropriate messages, so these will be available in time for the second stage of the study. Tufts and locally contracted researchers will collect information from program staff on their perception of the feasibility and impact of the change, and will interview beneficiaries to determine how they use the CSB and whether their use changes with the change in packaging/messaging. We may track the effect on intrahousehold sharing through self report of consumption among family members. This stage will last about six months, with data collection from beneficiaries conducted before and up to six months after the start of the intervention.

In addition to interviews and focus group discussions, we will collect samples of porridge as prepared in order to assess the proportion of oil, and we will conduct market observations to determine whether increased distribution of oil affects availability and price in the market, and whether market access affects beneficiary mothers' compliance with recommended preparation method. We will conduct a small number of in-home observations to observe beneficiary mothers' practices with respect to storage, preparation, and feeding of children, of which they might not be aware.

The key outcomes of the study are the proportion of oil in the CSB porridge as prepared, and the percent of beneficiary mothers who meet the standard for the oil : CSB ratio.

ELIGIBILITY:
All Beneficiary Mothers/Caretakers receiving supplementary food for their children at the selected FDPs implementing a program change or the control FDPs , are considered part of the subject pool. All beneficiaries will be receiving a program change (consistent with additional oil ration and education on preparation in Phase I, and repackaged CSB in Phase II) in the selected FDPs. Participation in individual interviews, focus group discussions, and observations constitutes subject participation.

Subject Categories

* Beneficiary Children that are part of the taste tests in preparation for Phase I
* Beneficiary Mothers/Caretakers that participate in interviews, focus group discussions, and in home observations
* Care Group Lead Mothers that participate in individual interviews and FGD
* Health Care Workers that participate in individual interviews
* PVO staff members that participate in individual interviews
* Store owners/Market Vendors that participate in individual interviews

Beneficiary Children (Children Under five years old,U5):

Inclusion Criteria:

* Child enrolled in Supplementary Feeding Program (SFP) to receive ration (CSB13 and FVO) from 1 of the 16 Food Distribution Points
* Child has an SFP ration card
* Subject's whose mother/caretaker or CSB preparer was contacted to participate in taste test FGD
* Subject's whose mother/caretaker is voluntarily willing to consent to their child's participation in taste tests

Exclusion Criteria:

- All children enrolled in the SFP in the selected program change FDPs are eligible

Beneficiary Mothers/Caretakers (Mothers/Caretakers of Children Under five years old,U5):

Inclusion Criteria:

* Beneficiary Mother/Caretaker enrolled in Supplementary Feeding Program (SFP) to receive ration (CSB13 and FVO) for her child from 1 of the 16 Food Distribution Points
* Beneficiary Child has an SFP ration card
* Beneficiary Mother/Caretaker has no age restrictions for inclusion (Note: Mothers/caretakers or CSB preparers will be asked to participate regardless of age and consented appropriately)
* Subject who is voluntarily willing to participate by signing the consent form (or if minor, adult is willing to sign on their behalf). Note: This should will only come after the subject has been educated on all that appertains to their her involvement in this study, the consent script read aloud for them and given the chance to make her own non-coerced, non-persuaded and autonomous decision.

Exclusion Criteria:

- Beneficiary Mothers/Caretakers who were interviewed once for this study will not be interviewed a second time during a later Phase of the study.

Care Group Lead Mothers

Inclusion Criteria:

* Lead mother who covers the catchment area of the selected 16 FDP's
* Lead mother has been present during the program change period
* Subject who is voluntarily willing to participate by signing the consent form

Exclusion Criteria:

- None

Health Care Workers (Health Surveillance Agents, Health Promoters, Resource Persons)

Inclusion Criteria:

* Health Care Workers serving within the catchment area for the 16 FDPs
* Health Care Worker has been present during the study period
* Subject who is voluntarily willing to participate by signing the consent form

Exclusion Criteria:

-None

PVO Staff Members

Inclusion Criteria:

* All staff members from Catholic Relief Services, Africare, Save the Children, Project Concern International (PCI)
* Subject who is voluntarily willing to participate by signing the consent form

Exclusion Criteria:

- PVO Staff members who joined too recently to have experience of the program change Store Owners/Market Vendor

Inclusion Criteria:

* Store owner/market vendor in study districts (i.e. Machinga, Balaka, Chiradzulu and Mulanje districts) who trades in the relevant products (food vendors)
* Subject who is voluntarily willing to participate by signing the consent form

Exclusion Criteria:

- Vendors who do not sell food.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 6811 (Actual)
Dates: Start 2013-07; Primary Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change in average percent of oil by volume in the porridge as prepared | Baseline (July 2013), Phase I (October 2013) 3 months, Phase II (January 2014) 6 months
  Having samples of prepared porridge taken from beneficiary mothers analyzed for percentage of oil content. This will allow us to know if the mothers are preparing the porridge in the appropriate ration of 100g CSB: 30g oil.

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice L Rogers, PhD, Principal Investigator — Tufts University
Locations (1):
- Blantyre, Malawi

REFERENCES:
- [Derived] Wilner L, Suri DJ, Langlois BK, Walton SM, Rogers BL. Effective delivery of social and behavior change communication through a Care Group model in a supplementary feeding program. J Health Popul Nutr. 2017 Sep 12;36(1):34. doi: 10.1186/s41043-017-0111-3. PMID 28899434